CLINICAL TRIAL: NCT02666248
Title: Long-term Follow-up of Subjects Exposed to Lentiviral-based CART-EGFRvIII Gene-modified Cellular Therapy Products in Cancer Studies
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC 11315, 823264
Record Dates: First submitted 2016-01-26; First posted 2016-01-28 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2019-01

CONDITIONS: Subjects Entering Into This Protocol Will be Followed for up to 15 Years After Initial CART-EGFRvIII Infusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This is a non-therapeutic, long-term follow-up (LTFU) study of subjects who have received retroviral-based gene therapy products in cancer studies. All subjects in this LTFU protocol have received lentiviral modified T cells engineered to express an anti-EGFRvIII scFv Chimeric Antigen Receptor (CAR).

DETAILED DESCRIPTION:
The primary objective of this study is to monitor adult subjects, who as participants of a clinical trial, received T cells modified by a lentiviral vector encoding a chimeric antigen receptor specific for EGFRvIII, for adverse events that may be associated with lentiviral vector gene transfer such as insertional oncogenesis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be enrolled into this destination protocol because they have received CART-EGFRvIII cells that were genetically modified with a lentiviral vector. All subjects who have participated in a lentiviral vector study under IND 15968 and have received CART-EGFRvIII cells will be asked to participate in this protocol.
* Subjects 18 years of age and older
* Subjects who have provided informed consent prior to their study participation.

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who have participated in a lentiviral vector study and have received CART-EGFRvIII cells.
Sampling Method: Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2016-05-23 (Actual); Primary Completion 2018-01-27 (Actual); Study Completion 2018-01-27 (Actual)

PRIMARY OUTCOMES:
Number of adverse events | 15 years

CONTACTS AND LOCATIONS:
Overall Officials: Donald O'Rourke, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (2):
- United States (2):
  - University of California, San Francisco, San Francisco, California
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania